CLINICAL TRIAL: NCT04612660
Title: Human Papillomavirus (HPV) and Cervical Cancer Intervention to Increase Cervical Cancer Screening for Underserved Asian Women
Brief Title: HPV Self-test to Increase Cervical Cancer Screening in Asian Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HPV Self-sampling
Record Dates: First submitted 2020-10-28; First posted 2020-11-03 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Physician Engagement; Patient Navigation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Specific Education and Dynamic Group (Experimental): 1. Motivational group education specifically focused on cervical cancer prevention;
  2. Dynamic group interaction and role play discussion sessions on the benefits of Self-Sample collection HPV testing and procedures;
  3. Engaging community bilingual physicians in cervical cancer screening and referral;
  4. Patient navigation assistance.
  Interventions: Behavioral: Education on cervical cancer prevetnion; Behavioral: Dynamic group interaction; Behavioral: Physician engagement; Behavioral: Patient Navigation
- General Health Education (Active Comparator): Comparison group participants received general health education focusing on healthy lifestyle, and prevention of disease through routine health examinations.
  Interventions: Behavioral: General Health Education

INTERVENTIONS:
Behavioral: Education on cervical cancer prevetnion — Motivational group education by trained bilingual community health educators (CHEs) on cervical cancer prevention
  Arms: Specific Education and Dynamic Group
Behavioral: Dynamic group interaction — Dynamic group interaction and role play discussion sessions on the benefits of Self-Sample collection HPV testing and procedures;
  Arms: Specific Education and Dynamic Group
Behavioral: Physician engagement — Engaging community bilingual physicians in cervical cancer screening and referral;
  Arms: Specific Education and Dynamic Group
Behavioral: Patient Navigation — Patient navigation assistance will be provided to participants who tested HPV positive for further diagnostic testing and treatment.
  Arms: Specific Education and Dynamic Group
Behavioral: General Health Education — general health education focusing on healthy lifestyle, and prevention of disease through routine health examinations.
  Arms: General Health Education

SUMMARY:
The study was to pilot test the feability of using HPV self-sampling testing to increase cervical cancer screening among under-served Asian women through engaging community-based organizations in the greater Philadelphia and New York City area, addressing a significant global cancer burden, the preventable infection-related cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

1. gender: female
2. age: 30-55
3. no current diagnosis of cervical cancer, and
4. have not participated in cervical cancer screening within the past 3 years.

Exclusion Criteria:

-

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 156 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
the change in the rate of cervical cancer screening | baseline, and 6-month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Grace Ma, PhD, Principal Investigator — Temple University
Locations (1):
- Center for Asian Health, Lewis Katz School of Medicine, Temple University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Ma GX, Zhu L, Zhai S, Lin TR, Tan Y, Johnson C, Fang CY, Belinson JL, Wang MQ. Empowering Low-Income Asian American Women to Conduct Human Papillomavirus Self-Sampling Test: A Community-Engaged and Culturally Tailored Intervention. Cancer Control. 2022 Jan-Dec;29:10732748221076813. doi: 10.1177/10732748221076813. PMID 35193408